CLINICAL TRIAL: NCT00237016
Title: Post Exposure Treatment With Doxycycline for the Prevention of Relapsing Fever
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: RF1
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Relapsing Fever, Tick-borne; Jarisch Herxheimer Reaction
MeSH Terms: conditions — Relapsing Fever

INTERVENTIONS:
Drug: doxycycline treatment

SUMMARY:
Abstract Background Tick-Borne Relapsing Fever (TBRF) is an acute febrile illness. In Israel, TBRF is caused by Borrelia persica and is transmitted by Ornithodoros tholozani ticks. We examined the safety and efficacy of a post exposure treatment policy to prevent TBRF.

Methods In a double blind, placebo controlled trial 93 healthy volunteers with suspected tick exposure (51 with bite signs and 42 contacts) were randomly assigned to receive either Doxycycline (200 mg for the first day and 100mg/d for 4 days) or placebo, approximately 2 days after contact. Blood smears were examined for Borrelia at inclusion and during fever rise. Serology for Lyme disease cross- reactivity and PCR for Borrelia GlpQ gene were also performed. Cases of TBRF were defined as subjects having fever and a positive blood smear.

ELIGIBILITY:
Inclusion Criteria:

* suspected exposure to tick-borne relapsing fever
* after returning from field exercise in a tick-borne relapsing fever infected area
* having a tick bite or staying in field in close proximity to a subject with tick bite sign

Exclusion Criteria:

* known sensitivity to tetracycline or doxycycline
* febrile illness on recruitment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140
Dates: Start 2002-04; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Overall Officials: Tal Hasin, MD, Principal Investigator — Medical corps, Israel Defence Forces
Locations (1):
- Israel Defence Forces, Tel Litwinsky, Israel

REFERENCES:
- [Background] Nadelman RB, Nowakowski J, Fish D, Falco RC, Freeman K, McKenna D, Welch P, Marcus R, Aguero-Rosenfeld ME, Dennis DT, Wormser GP; Tick Bite Study Group. Prophylaxis with single-dose doxycycline for the prevention of Lyme disease after an Ixodes scapularis tick bite. N Engl J Med. 2001 Jul 12;345(2):79-84. doi: 10.1056/NEJM200107123450201. PMID 11450675
- [Derived] Hasin T, Davidovitch N, Cohen R, Dagan T, Romem A, Orr N, Klement E, Lubezky N, Kayouf R, Sela T, Keller N, Derazne E, Halperin T, Yavzori M, Grotto I, Cohen D. Postexposure treatment with doxycycline for the prevention of tick-borne relapsing fever. N Engl J Med. 2006 Jul 13;355(2):148-55. doi: 10.1056/NEJMoa053884. PMID 16837678